CLINICAL TRIAL: NCT00347594
Title: A Clinical Evaluation of the Next Generation Diagnostic Instrument (NGDI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GVC2-03-052
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Corneal surface topography; Ocular aberrations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Next Generation Diagnostic Instrument (Experimental): Next Generation Diagnostic Instrument (NGDI)
  Interventions: Device: Next Generation Diagnostic Instrument (NGDI)
- Zyoptix Diagnostic Workstation (Active Comparator): Zyoptix Diagnostic Workstation (ZDW)
  Interventions: Device: Zyoptix Diagnostic Workstation (ZDW)

INTERVENTIONS:
Device: Next Generation Diagnostic Instrument (NGDI) — Measurement of the aberrations, corneal surface topography, and pachymetry of normal human eyes
  Arms: Next Generation Diagnostic Instrument
Device: Zyoptix Diagnostic Workstation (ZDW) — Measurement of the aberrations, corneal surface topography, and pachymetry of normal human eyes
  Arms: Zyoptix Diagnostic Workstation

SUMMARY:
The purpose of this study is to measure the aberrations, corneal surface topography and pachymetry of normal human eyes with the NGDI.

ELIGIBILITY:
Inclusion Criteria:

* +10.00D to -20.00D of absolute spherical ametropia
* Must be part of the Bausch & Lomb research clinic
* Snellen visual acuity must be correctable to 20/25

Exclusion Criteria:

* No more than -6.00D of refractive astigmatism

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Measurement of aberrations with the NGDI and the Zywave II. | Single visit

SECONDARY OUTCOMES:
Measurement of corneal topography and pachymetry with the NGDI and the Orbscan IIz. | Single visit

CONTACTS AND LOCATIONS:
Overall Officials: Michele Lagana, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States